CLINICAL TRIAL: NCT01611142
Title: Open-Label, Multi-Center, Phase 2 Study of Anti-CCR4 Monoclonal Antibody KW-0761 (Mogamulizumab) in Subjects With Previously Treated Peripheral T-cell Lymphoma (PTCL)
Brief Title: Study of KW-0761 (Mogamulizumab) in Subjects With Previously Treated Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTOCOL 0761-007
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Monoclonal antibody; Peripheral T-cell Lymphoma; cancer; hematologic malignancy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Neoplasms; Hematologic Neoplasms | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KW-0761 (Experimental)
  Interventions: Biological: KW-0761 (mogamulizumab)

INTERVENTIONS:
Biological: KW-0761 (mogamulizumab) — 1 mg/kg administered intravenously weekly x 4 then every other week until progression
  Other Names: mogamulizumab; POTELIGEO®

SUMMARY:
The primary objective of this study is to determine the overall response rate of KW-0761 for the treatment of patients with relapsed or refractory PTCL. KW-0761 targets CCR4. CCR4 is the receptor for macrophage derived chemokines MDC/CCL22 and TARC/CCL17. Chemokines are considered to play a role both in the recruitment of immune and inflammatory cells for anti-tumor response and in the selective homing of neoplastic B and T cells.

DETAILED DESCRIPTION:
PTCL is a rare and heterogeneous disease that remains difficult to diagnose and treat. In the majority of PTCL subtypes, patients are of older age (>60 years) and present with advanced stage disease.With the exception of the ALCL-ALK-positive subtype that responds well to CHOP combined chemotherapy, most PTCL subtypes become refractory even to aggressive chemotherapy regimens or relapse. Overall survival of PTCL patients is poor compared with that of aggressive B-cell lymphomas.Thus, novel and effective therapies are needed.KW-0761(mogamulizumab) is a defucosylated, humanized, IgG1 mAb with enhanced antibody dependent cellular cytotoxicity (ADCC)that binds to CCR4, a molecule that is suggested to be significantly involved in patients with PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of enrollment;
2. Histologically confirmed diagnosis of PTCL as specified below:

   * PTCL-NOS
   * Angioimmunoblastic T-cell lymphoma
   * Anaplastic large cell lymphoma, ALK-positive
   * Anaplastic large cell lymphoma, ALK-negative
   * Transformed mycosis fungoides
3. Failed or intolerant of at least one prior systemic anticancer therapy;
4. ECOG performance status score of ≤ 2 at study entry;
5. At least one site of disease measurable in two dimensions by computed tomography (CT);
6. Subjects who are positive for CCR4 by immunohistochemistry;
7. Resolution of all clinically significant toxic effects of prior cancer therapy to grade ≤1 (NCI-CTCAE, v.4.0);
8. Adequate hematological hepatic and renal function.

Exclusion Criteria:

1. Subject with the following PTCL diagnoses are excluded;

   * Precursor T/NK neoplasms
   * Adult T-cell leukemia-lymphoma
   * T-cell prolymphocytic leukemia
   * T-cell large granular lymphocytic leukemia
   * Aggressive NK-cell leukemia
   * Systemic EBV-positive T-cell lymphoproliferative disorder of childhood
   * Hydroa vacciniforme-like lymphoma
   * Mycosis fungoides, other than transformed mycosis fungoides
   * Sezary Syndrome
   * Primary cutaneous CD30+ disorders: Anaplastic large cell lymphoma and lymphatoid papulosis
   * Primary cutaneous CD8+ aggressive epidermotropic cytoxic T-cell lymphoma
   * Primary cutaneous CD4+ small/medium T-cell lymphoma
   * Primary cutaneous gamma-delta T-cell lymphoma
   * Extranodal NK/T T-cell lymphoma-nasal type
   * Enteropathy-associated T-cell lymphoma
   * Hepatosplenic T-cell lymphoma
   * Subcutaneous panniculitis -like T-cell lymphoma
   * Chronic lymphoproliferative disorder of NK cells
2. Have had an invasive solid tumor malignancy in the past five years except non-melanoma skin cancers, melanoma in situ, cervical carcinoma in situ, ductal/lobular carcinoma in situ of the breast, or localized prostate cancer with a current PSA of ≤ 0.1 ng/ml who is currently without evidence of disease;
3. Relapsed less than 75 days of autologous stem cell transplant;
4. History of allogeneic stem cell transplant;
5. Evidence of central nervous system (CNS) metastasis;
6. Psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit compliance with study requirements;
7. Subjects with a history of moderate or severe psoriasis or with psoriasis associated with systemic symptoms e.g. arthropathy), or with a 1st degree relative with history of psoriasis that required medical intervention;
8. Significant uncontrolled intercurrent illness;
9. Known or tests positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C;
10. Active herpes simplex or herpes zoster;
11. Experienced allergic reactions to monoclonal antibodies or other therapeutic proteins;
12. Known active autoimmune disease will be excluded (For example: Grave's disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease);
13. Is pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or lactating; Prohibited Therapies and/or Medications
14. Prior treatment with KW-0761;
15. Initiation of treatment with systemic steroids while on study is only permitted for acute and brief complications of underlying disease (e.g., hypercalcemia) or for treatment related side effects;
16. Initiation of treatment with topical steroids while on study is not permitted except to treat an acute rash;
17. Have had anti-neoplastic chemotherapy, radiation, immunotherapy, or investigational medications within 4 weeks of screening visit;
18. Subjects on any immunomodulatory drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, M.D., PhD, Principal Investigator — Universita di Bologna
Locations (15):
- Aarhus University Hospital, Aarhus, Denmark
- France (5):
  - CHU Henri Mondor, Créteil
  - CHRU Lille, Lille
  - Hopital Saint-Louis, Paris
  - Centre Hospitaliser de Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
- Università di Bologna, Bologna, Italy
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
- Spain (3):
  - Institut Catalá D'Oncologia, Hospital Duran y Reynals, Barcelona
  - Hospital Univesitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - Guy's Hospital, London
  - Christie Hospital, Manchester
  - Cancer Research UK Centre/Southhampton General Hospital, SouthHampton

REFERENCES:
- [Derived] Zinzani PL, Karlin L, Radford J, Caballero D, Fields P, Chamuleau ME, d'Amore F, Haioun C, Thieblemont C, Gonzalez-Barca E, Garcia CG, Johnson PW, van Imhoff GW, Ng T, Dwyer K, Morschhauser F. European phase II study of mogamulizumab, an anti-CCR4 monoclonal antibody, in relapsed/refractory peripheral T-cell lymphoma. Haematologica. 2016 Oct;101(10):e407-e410. doi: 10.3324/haematol.2016.146977. Epub 2016 Jul 14. No abstract available. PMID 27418646